CLINICAL TRIAL: NCT03261063
Title: China Evera MRI® Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: China Evera
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evera Implanted Group (Experimental)
  Interventions: Device: Evera MRI ICD System

INTERVENTIONS:
Device: Evera MRI ICD System — Subjects are implanted with Evera MRI ICD System and exposed to MRI environment per study requirements

SUMMARY:
The study is a prospective, single arm, non-blinded, multi-site study conducted in mainland China.

DETAILED DESCRIPTION:
The purpose of the China Evera MRI® study is to confirm safety of the Evera MRI ICD System in the clinical MRI (Magnetic Resonance Imaging) environment when subjects receive MRI scans up to 2W/kg Specific Absorption Rate (SAR) without positioning restrictions (MRI scans may occur anywhere on the body). Long-term device effects, such as long-term lead integrity, will not be assessed in the China Evera MRI® study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are indicated for implantation of an ICD at the time of study enrollment.
* Subjects who are able to undergo a pectoral implant.
* Subjects who are able and willing to undergo elective MRI scanning without sedation , .
* Subjects who are geographically stable and available for follow-up at the study site for the length of the study.
* Subjects who are at least 18 years of age (or older, if required by local law).

Exclusion Criteria:

* Subjects with a history of significant tricuspid valvular disease that precludes the ability to place the RV lead. .
* Subjects who may be contraindicated to the dexamethasone sodium phosphate and/or dexamethasone acetate.
* Subjects who require a legally authorized representative to obtain informed consent.
* Subjects with abandoned or capped leads.
* Subjects who require an indicated MRI scan, other than those specifically described in the China Evera MRI® study, before the one-month post-MRI follow-up (approximately 4 months post-implant).
* Subjects with a non-MRI compatible device (such as neurostimulators) or material implant (e.g., non-MRI compatible sternal wires, neurostimulators, biostimulators, metals or alloys).
* Subjects with medical conditions that preclude the testing required by the CIP or limit study participation.
* Subjects who are enrolled or intend to participate in another clinical trial (of an investigational drug or device, new indication for an approved drug or device, or requirement of additional testing beyond standard clinical practice) during the China Evera MRI® study. Co-enrollment in concurrent trials is only allowed when documented pre-approval is obtained from the Medtronic study manager.
* Female patient who is pregnant, or of childbearing potential and not on a reliable form of birth control. Women of childbearing potential are required to have a negative pregnancy test within seven (7) days prior to device implant
* Subjects with exclusion criteria required by local law (e.g., age, breastfeeding).
* Subjects who are diagnosed with terminal disease with life expectancy less than 4 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
The proportion of successful MRI scans | 1 Month Follow up visit after MRI Scan Visit
  To summarize the MRI-related event rate within 30 days post-MRI in patients implanted with an Evera MRI device.

SECONDARY OUTCOMES:
The effectiveness of the Evera MRI device post-MRI. | Pre-MRI scan, immediately post MRI scan, 1-week and 1-month post MRI scan.
  The effectiveness of the Evera MRI device will be measured by the following parameters
  1. Atrial pacing capture threshold (only for dual chamber devices)
  2. Atrial sensing amplitude (only for dual chamber devices)
  3. Ventricular pacing capture threshold
  4. Ventricular sensing amplitude These parameters will be measured pre-MRI scan, immediately post MRI scan, 1-week and 1-month post MRI scan.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Hua Xi Hospital (West China Hospital), Chengdu, Sichuan